CLINICAL TRIAL: NCT01375127
Title: An Observational Study To Collect Follow-up Clinical Data From Kidney Transplant Recipients Who Received Tofacitinib (CP-690,550) In Completed Phase 2 Studies
Brief Title: Collection of Follow-up Data From CP-690,550-treated Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921053
Record Dates: First submitted 2011-06-13; First posted 2011-06-17 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-09

CONDITIONS: Kidney Transplantation
Keywords: Observational; clinical follow-up data
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects from Study A3921009
  Interventions: Drug: Tofacitinib
- Subjects from Study A3921030
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Subjects who previously took 15 mg BID or 30 mg BID
  Groups: Subjects from Study A3921009
Drug: Tofacitinib — Subjects who previously took 15 mg BID for 3 months then 10 mg BID, or 15 mg BID for 6 months then 10 mg BID
  Groups: Subjects from Study A3921030

SUMMARY:
This is an observational study designed to collect follow-up clinical date on subjects who were treated with tofacitinib in 2 completed Phase 2 studies who either discontinued treatment prematurely or did not elect to enroll in long-term extension studies.

DETAILED DESCRIPTION:
Subjects are identified based on whether they received tofacitinib in 2 completed Phase 2 studies who either discontinued treatment prematurely or who did not elect to enroll in long-term extension studies. Subjects are pre-identified

ELIGIBILITY:
Inclusion Criteria:

* Subjects have discontinued tofacitinib prior to the planned treatment duration in 2 completed Phase 2 studies; or have not enrolled in long-term extension studies.

Exclusion Criteria:

* No other subjects are eligible for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received treatment with tofacitinib in 2 completed Phase 2 studies who either discontinued treatment prematurely or who did not elect to enroll in long-term extension studies.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (19):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Springfiled, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Valhalla, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Richmond, Virginia
- Australia (5):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
- Pfizer Investigational Site, Anderlecht, Belgium
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Edmonton, Alberta, Canada
- Pfizer Investigational Site, Praha 4 - Krc, Czechia
- France (3):
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Toulouse
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Hamburg
- Pfizer Investigational Site, Roma, Italy
- Pfizer Investigational Site, Rotterdam, Netherlands
- Pfizer Investigational Site, Oslo, Norway
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921053&StudyName=Collection%20of%20follow-up%20data%20from%20CP-690%2C550-treated%20kidney%20transplant%20recipients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who discontinued tofacitinib prior to the end of the planned treatment duration, or did not enroll in long-term extension studies after completing tofacitinib treatment in Phase 2a study A3921009 (NCT00106639) and Phase 2b study A3921030 (NCT00483756) were enrolled in this study.
Groups:
- Tofacitinib 10 mg (Pre-amendment 1, Study A3921030): Participants who received tofacitinib 10 milligram (mg) tablet orally twice daily during study A3921030 (NCT00483756) pre-amendment 1 were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of post-transplant lymphoproliferative disease (PTLD), central nervous system (CNS) infection, graft failure and death (if any).
- Tofacitinib 15 mg (Pre-amendment 1, Study A3921030): Participants who received tofacitinib 15 mg tablet orally twice daily during study A3921030 (NCT00483756) pre-amendment 1 were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of PTLD, CNS infection, graft failure and death (if any).
- Tofacitinib 15 mg (Study A3921030, Month 1 to 6): Participants who received tofacitinib 15 mg tablet orally twice daily for Month 1 to 6 during study A3921030 (NCT00483756) were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of PTLD, CNS infection, graft failure and death (if any).
- Tofacitinib 15 mg (Study A3921030, Month 1 to 3): Participants who received tofacitinib 15 mg tablet orally twice daily for Month 1 to 3 during study A3921030 (NCT00483756) were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of PTLD, CNS infection, graft failure and death (if any).
- Tofacitinib 15 mg (Study A3921009): Participants who received tofacitinib 15 mg tablet orally twice daily up to Month 6 during study A3921009 (NCT00106639) were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of PTLD, CNS infection, graft failure and death (if any).
- Tofacitinib 30 mg (Study A3921009): Participants who received tofacitinib 30 mg tablet orally twice daily up to Month 6 during study A3921009 (NCT00106639) were followed-up through 12 months after the last dose of tofacitinib to evaluate occurrence of PTLD, CNS infection, graft failure and death (if any).
Period: Overall Study
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Started | 1 | 1 | 40 | 33 | 5 | 3
Completed | 1 | 1 | 40 | 33 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009) | Total
Number analyzed (Participants) | 1 | 1 | 40 | 33 | 5 | 3 | 83
Age Continuous [Mean (Standard Deviation); unit: years] | 67.0 | 26.0 | 46.8 (13.2) | 45.3 (13.1) | 46.8 (8.5) | 36.7 (3.1) | 45.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 7 | 6 | 4 | 0 | 17
  Male | 1 | 1 | 33 | 27 | 1 | 3 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Outcome of Post Transplant Lymphoproliferative Disease (PTLD)
Description: All lymphoproliferative disorders diagnosed locally as PTLD based on histopathology were reported.
Time Frame: Baseline through Month 12
Population: Safety analysis included all eligible participants who had provided an informed consent for this study.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Number analyzed (Participants) | 1 | 1 | 40 | 33 | 5 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Central Nervous System (CNS) Infection
Description: Participants with CNS infection involving the brain or spinal cord, within 12 months after the last dose of tofacitinib were reported.
Time Frame: Baseline through Month 12
Population: Safety analysis included all eligible participants who had provided an informed consent for this study.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Number analyzed (Participants) | 1 | 1 | 40 | 33 | 5 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Graft Failure
Description: Graft failure which occurred within 12 months after the last dose of tofacitinib was reported. Graft failure was defined as graft nephrectomy, re-transplantation, or return to dialysis for greater than or equal to (>=) 6 consecutive weeks.
Time Frame: Baseline through Month 12
Population: Safety analysis included all eligible participants who had provided an informed consent for this study.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Number analyzed (Participants) | 1 | 1 | 40 | 33 | 5 | 3
participants | 0 | 0 | 2 | 3 | 0 | 0

4. Primary Outcome: Number of Participants Who Died
Time Frame: Baseline through Month 12
Population: Safety analysis included all eligible participants who had provided an informed consent for this study.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Number analyzed (Participants) | 1 | 1 | 40 | 33 | 5 | 3
participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Data collection was limited to clinical outcome of PTLD, CNS infection, graft failure, or death. Clinical outcomes were to be reported as serious adverse event (SAE) if they met pre-defined SAE criteria and had causal relationship to tofacitinib. Non-SAEs were not planned to be reported.
Arm/Group | Tofacitinib 10 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Pre-amendment 1, Study A3921030) | Tofacitinib 15 mg (Study A3921030, Month 1 to 6) | Tofacitinib 15 mg (Study A3921030, Month 1 to 3) | Tofacitinib 15 mg (Study A3921009) | Tofacitinib 30 mg (Study A3921009)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/40 | 0/33 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.